CLINICAL TRIAL: NCT07066618
Title: Effects of Meal Energy Density on Anthropometric Measurements, Some Metabolic Parameters, And Subjective Appetite in Women
Brief Title: Effects of Meal Energy Density on Body Measures and Metabolism in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melike Nur Eroğlu (Other)
Responsible Party: Sponsor-Investigator, Melike Nur Eroğlu, Lecturer, Sakarya Applied Sciences University
Organization: Sakarya Applied Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BASKENT-MEALTIME-2023
Record Dates: First submitted 2025-06-15; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Overweight; Appetite Regulation; Meal Timing; Circadian Rhythm; Metabolic Health
Keywords: circadian rhythm; appetite; Meal Timing; obesity; Glucose Metabolism
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breakfast Group (BG) (Experimental)
  Interventions: Behavioral: Breakfast-Loaded Hypocaloric Diet
- Dinner Group (DG) (Experimental)
  Interventions: Behavioral: Dinner-Loaded Hypocaloric Diet

INTERVENTIONS:
Behavioral: Breakfast-Loaded Hypocaloric Diet — Participants in this group consumed a hypocaloric diet in which 50% of daily energy intake was provided at breakfast, 35% at lunch, and 15% at dinner. Meal times were standardized as follows: breakfast (7:00-9:00), lunch (12:00-14:00), and dinner (18:00-20:00). The diet was individually tailored and provided 20% fewer calories than the participants' total energy expenditure. Macronutrient distribution followed recommended guidelines: 45-60% carbohydrates, 10-20% protein, and 20-35% fat.
  Arms: Breakfast Group (BG)
Behavioral: Dinner-Loaded Hypocaloric Diet — Participants in this group consumed a hypocaloric diet in which 15% of daily energy intake was provided at breakfast, 35% at lunch, and 50% at dinner. Meal times were standardized as follows: breakfast (7:00-9:00), lunch (12:00-14:00), and dinner (18:00-20:00). The diet was individually tailored and provided 20% fewer calories than the participants' total energy expenditure. Macronutrient distribution followed recommended guidelines: 45-60% carbohydrates, 10-20% protein, and 20-35% fat.
  Arms: Dinner Group (DG)

SUMMARY:
This study investigates whether the timing of energy intake during the day-specifically consuming more calories at breakfast or at dinner-affects body measurements, blood sugar levels, cholesterol, and feelings of hunger in women who are overweight or obese.

A total of 28 women participated in the study and were randomly assigned to one of two diet plans: one group consumed half of their daily calories at breakfast, while the other consumed them at dinner. Both groups followed a calorie-restricted diet for six weeks.

The goal of this research is to understand whether eating more in the morning rather than in the evening leads to better outcomes for weight control and metabolic health. Findings from this study may help health professionals make more effective meal timing recommendations for weight loss and improving blood sugar regulation.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-45
* BMI ≥25 kg/m²
* Regular menstrual cycle
* No chronic disease or medication use
* PSQI ≤5 (Good sleep quality)

Exclusion Criteria:

* Pregnancy or lactation
* Gastrointestinal or metabolic disorders
* Shift workers, sleep disorders
* Medication affecting metabolism
* Weight change >4.5 kg in last 6 months

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Change in fasting blood glucose | Baseline to Week 6

SECONDARY OUTCOMES:
Change in hip circumference | Baseline to Week 6
Change in HDL cholesterol | Baseline to Week 6
Change in HbA1c | Baseline to Week 6

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University of Applied Sciences, Faculty of Sport Sciences, Exercise and Sports Sciences Education, Application and Research Centre, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Informed Consent Form (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT07066618/ICF_000.pdf